CLINICAL TRIAL: NCT02082990
Title: A Randomised Controlled Non-inferiority Trial of Primary Care-based Facilitated Access to a Web Based Brief Intervention to Reduce Alcohol Consumption (EFAR-Spain)
Brief Title: Primary Care-based Facilitated Access to a Web Based Brief Intervention to Reduce Alcohol Consumption
Acronym: EFAR-Spain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: August Pi Sunyer Biomedical Research Institute (Other); Fundacion Clinic per a la Recerca Biomédica (Other); Program on Substance Abuse, Public Health Agency, Government of Catalonia (Unknown); University College, London (Other); Instituto de Salud Carlos III (Other Government); European Union (Other)
Responsible Party: Principal Investigator, Antoni Gual, Senior Consultor, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI042924
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Hazardous Drinking
Keywords: Alcohol-related disorders; Alcohol Drinking; e-health; Alcohol Use Disorder Test; Quality of Life
MeSH Terms: conditions — Alcohol-Related Disorders; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Face-to-Face Brief Intervention Group (Active Comparator): One face-to-face Brief Intervention which is provided by General Practitioner or Nurse
  Interventions: Behavioral: Face-to-Face Brief Intervention
- Online Brief Intervention Group (Experimental): Primary care-based facilitated access to an alcohol reduction website (Brief Intervention)
  Interventions: Behavioral: Online Brief Intervention

INTERVENTIONS:
Behavioral: Face-to-Face Brief Intervention — One face-to-face Brief Intervention which is provided by General Practitioner or Nurse
  Arms: Face-to-Face Brief Intervention Group
Behavioral: Online Brief Intervention — Primary care-based facilitated access to an alcohol reduction website (Brief Intervention)
  Arms: Online Brief Intervention Group

SUMMARY:
Brief Interventions (BIs) for risky drinkers are an effective tool in primary care. Lack of time in daily practice has been identified as a barrier for the wide implementation of BI. There is growing evidence that e-health tools such as web based BIs can be an efficient alternative to standard face-to-face BIs and save time to general practitioners (GP).

The main aim of this study is to test non-inferiority of a web based BI for risky drinkers against a traditional face to face BI delivered by a general practitioner. We have designed a randomised controlled non-inferiority trial comparing both interventions, to be performed in primary care health centres in Catalonia, Spain.

Adults attending in primary care centres and willing to participate, will be invited to fill the short Alcohol Use Disorders Identification Test (AUDIT-C) in a specific website. Those screening positive and who accept to share the baseline data with their GP will be invited to an online assessment of their drinking and randomized to a standard BI with their GP or to the online BI.

Follow-up assessment will be conducted online at months 3 and 12, using the full Alcohol Use Disorder Identification Test (AUDIT) and the quality of life questionnaire (D5-EQD5). The main outcome will be the proportion of risky drinkers according to the AUDIT. Assuming a 30% reduction in the proportion of risky drinkers in the control group (classroom), allowing for an overall attrition of 10% of patients in the trial and non-inferiority assessed against a specified margin of 10%, it is estimated that 500 patients would be required in each group to give the test a 90% power (1-β) to reject the null hypothesis.

DETAILED DESCRIPTION:
Trial design: A randomised non-inferiority controlled trial in primary care comparing facilitated access to a website for risky drinkers against a standard face-to-face BI. With the exception of the non-experimental intervention, all components of the study will be administered online to patients. Patients will be actively encouraged by their PHCP to access the application, which is available on the website of the programme 'Alcohol y Salud' (http:// www.alcoholysalud.cat), and will be provided with a unique registration code. The trial website is a Spanish adaptation of the English version of http://www.DownYourDrink.org.uk (DYD) developed in the UK, which includes modules for all the key trial components including screening, consent, assessment, randomisation and follow-up. It also incorporates the alcohol reduction website for the patients in the experimental group. The site has been adapted from the http://www.DownYourDrink.org.uk website developed for the DYD-RCT (randomised controlled trial).14 Details of DYD and the psychological theory that underpinned its development have been reported elsewhere. 21 Country-specific information such as recommended guidelines for alcohol intake, definitions of standard drinks and alcohol-related laws will be included. The website also incorporates a menu-driven facility to enable PHCP to customise automated messages to patients, for example, by adding photographs and pre-recorded messages. The personalised messages will appear to each patient using the log-in code provided by that practitioner.

Practitioner recruitment, training and incentives:

Recruitment will be based on the XaROH network. A 3 h seminar on new technologies, and EI and BI, introducing the trial, will be offered to all members of the XaROH, and those attending will be invited to sign up for the trial. In addition, several advertisements will be posted on the 'Beveu Menys' platform offering participation in the trial. In selecting practices, preference will be given to those with at least 5000 registered patients. Those practices that are selected as participants will be required to undergo a 1-day training programme. The training has four steps: (1) introduction to trial; (2) familiarisation with website; (3) update about EI and BI; and (4) practice in EI and BI (role-playing). Finally, participants will be encouraged to use the website and to tailor-make patient messages. Participating PHCPs will receive a financial incentive of €20 per patient recruited to the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or over attended in primary care during the study period
* AUDIT-C 4 or above for women and 5 or above for men (in online screening)

Exclusion Criteria:

* Severe psychiatric disorders
* Serious visual impairment
* Terminal illness
* To have inadequate command of the Spanish or Catalan language
* AUDIT ≥ 18 in baseline assessment.

Excluded patients will be referred to GPs to consider other interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of risky drinkers according to the Alcohol Use Disorder Identification Test (AUDIT) | At month 3 after the randomisation
  % of patients with > 7 scoring in AUDIT (month 3)

SECONDARY OUTCOMES:
Proportion of risky drinkers according to the Alcohol Use Disorder Identification Test (AUDIT) | at month 12 after the randomisation
  % of patients with > 7 scoring in AUDIT (month 12)
Quality of life EQ-5D-3L questionnaire | at month 3 and 12 after the randomisation
  Increasing of QoL according to EQ5D53L

OTHER OUTCOMES:
Implementation | at month 3 after the randomisation
  Proportion of Brief Interventions carried out among the subjects who are positively screened

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gual, MD. PhD, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- Primary Care Centres of Institut Català de la Salut, Multiple Locations, Catalonia, Spain

REFERENCES:
- [Derived] Lopez-Pelayo H, Wallace P, Segura L, Miquel L, Diaz E, Teixido L, Baena B, Struzzo P, Palacio-Vieira J, Casajuana C, Colom J, Gual A. A randomised controlled non-inferiority trial of primary care-based facilitated access to an alcohol reduction website (EFAR Spain): the study protocol. BMJ Open. 2014 Dec 31;4(12):e007130. doi: 10.1136/bmjopen-2014-007130. PMID 25552616
- See also: BMJ Open: A randomised controlled non-inferiority trial of primary care-based facilitated access to an alcohol reduction website (EFAR Spain): the study protocol — http://bmjopen.bmj.com/content/4/12/e007130